CLINICAL TRIAL: NCT02470312
Title: MediGuide Registry
Status: Terminated | Type: Observational
Why Stopped: Existing trials demonstrate reduction in fluoroscopy with MediGuide
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 10051
Record Dates: First submitted 2015-04-28; First posted 2015-06-12 (Estimated); Results first posted 2019-01-11 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Heart Failure; Cardiac Arrhythmia
Keywords: utility of MediGuide system; CRT; EP
MeSH Terms: conditions — Heart Failure; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CRT: Patients who are undergoing CRT implantation utilizing MediGuide system and tools
  Interventions: Procedure: CRT implantation; Device: MediGuide
- EP: Patients who are undergoing ablation procedures for Atrial Fibrillation, Atrial Flutter, and Ventricular Tachycardia utilizing MediGuide system and tools
  Interventions: Device: MediGuide; Procedure: EP

INTERVENTIONS:
Procedure: CRT implantation — It is a novel 3D electromagnetic navigation system (MediGuide™) that is capable of non-fluoroscopic navigation of sensor-enabled tools in the x-ray environment
  Groups: CRT
Device: MediGuide
Procedure: EP
  Groups: EP

SUMMARY:
The goal of this registry/observational study is to collect data on the clinical utility of MediGuide™ system in cardiac resynchronization therapy (CRT) implantation and electrophysiology (EP) procedures.

DETAILED DESCRIPTION:
The intent of this worldwide registry/observational study is to understand the utility of the MediGuide™ technology in real world clinical practice during CRT implantation and study-specific-EP procedures. The study should provide an understanding of the effect of MediGuide™ technology on:

* The amount of fluoroscopy time and the radiation exposure
* Total procedure time
* Peri-procedural clinical event rate

Additionally, this study will address the following

* Identification of procedural challenges which may aid in developing future MediGuide tools
* Evaluation of newly available MediGuide tools during the study
* Correlation between MediGuide operator experience and the radiation exposure amount and time

ELIGIBILITY:
Inclusion Criteria:

* Anybody coming for CRT or EP procedure utilizing MediGuide system and tools

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CRT Group All patients from participating sites who are indicated for a CRT-D/P device implant, including an upgrade with a new left ventricular (LV) lead implant and are implanted with St. Jude Medical pulse generators and willing to provide written Informed Consent can be enrolled in this study. Patients can be implanted with non-St. Jude Medical leads
  EP Group All patients from participating sites who are indicated for an atrial fibrillation, atrial flutter or ventricular tachycardia (VT) ablation procedure for which market approved MediGuide™-enabled ablation catheter is available and willing to provide written Informed Consent can be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 578 (Actual)
Dates: Start 2015-08-18 (Actual); Primary Completion 2017-02-10 (Actual); Study Completion 2018-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Ruffner, PhD, Study Director — Abbott
Locations (16):
- United States (6):
  - John C Lincoln North Mountain Hospital, Phoenix, Arizona
  - Athens Regional Medical Center, Athens, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Central Baptist Hospital, Lexington, Kentucky
  - North Texas Heart Center, Dallas, Texas
  - Memorial Hermann Southwest Hospital, Houston, Texas
- St. Andrews War Memorial Hospital, East Brisbane, Australia
- A. ö. Krankenhaus der Elisabethinen Linz, Linz, Austria
- Institut de Cardiologie de Montreal, Montreal, Canada
- Tartu University Hospital, Tartu, Estonia
- Germany (4):
  - Klinikum Inglostadt, Ingolstadt
  - Herzzentrum Leipzig, Leipzig
  - Deutsches Herzzentrum München des Freistaates Bayern, München
  - Kliniken Villingen-Schwenningen, Villingen-Schwenningen
- Leiden University Medical Center, Leiden, Netherlands
- Clinica Universitaria de Navarra, Pamplona, Spain

RESULTS

PARTICIPANT FLOW:
Groups:
- CRT Group: All subjects willing to provide written informed consent from participating sites, who were indicated for a CRT-D/P device implant (including an upgrade with a new LV lead) and were implanted with a SJM pulse generator, utilizing the MediGuide system and tools, were enrolled in this registry. Subjects could be implanted with non-SJM leads.
- EP Group: All subjects willing to provide written informed consent from participating sites, who were undergoing ablation procedures for atrial fibrillation, atrial flutter and ventricular tachycardia, utilizing the MediGuide system and tools, were enrolled in this registry.
Period: Overall Study
Arm/Group | CRT Group | EP Group
Started | 147 | 431
Completed | 142 | 419
Not Completed | 5 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CRT Group | EP Group | Total
Number analyzed (Participants) | 147 | 431 | 578
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.8 (10.3) | 62.5 (12.5) | 64.6 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 129 | 171
  Male | 105 | 302 | 407
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 36 | 28 | 64
  Austria | 0 | 11 | 11
  Netherlands | 0 | 16 | 16
  United States | 72 | 90 | 162
  Australia | 0 | 26 | 26
  Germany | 7 | 132 | 139
  Estonia | 25 | 27 | 52
  Spain | 0 | 46 | 46
  Italy | 2 | 3 | 5
  Taiwan | 0 | 10 | 10
NYHA classification [Count of Participants; unit: Participants] — The New York Heart Association (NYHA) Classification provides a simple way of classifying the extent of heart failure. It classifies patients in one of four categories based on their limitations during physical activity; the limitations/symptoms are in regards to normal breathing and varying degrees in shortness of breath and or angina pain.
  NYHA I: - No symptoms and no limitation in ordinary physical activity NYHA II: Mild symptoms / slight limitation during ordinary activity. NYHA III: Marked limitation in activity due to symptoms NYHA IV: Severe limitations, even while at rest.
  Participants
    NYHA I | 2 | 120 | 122
    NYHA II | 45 | 102 | 147
    NYHA III | 66 | 27 | 93
    NYHA IV | 2 | 4 | 6
    NOT AVAILABLE | 32 | 178 | 210
LEFT VENTRICULAR EJECTION FRACTION [Mean (Standard Deviation); unit: PERCENTAGE] | 29.1 (10.2) | 55.1 (11.5) | 48.0 (16.1)

OUTCOME MEASURES:

1. Primary Outcome: Amount of Fluoroscopy Time
Description: Amount of fluoroscopy time during CRT implant or EP procedure
Time Frame: Expected time frame is day 1 of the study
Measure: Mean (Standard Deviation); unit: MINUTES
Arm/Group | CRT Group | EP Group
Number analyzed (Participants) | 142 | 419
MINUTES | 9.5 (8.0) | 6.0 (9.9)

2. Primary Outcome: Periprocedural Adverse Event
Description: Adverse event until patients are discharged from the site center
Time Frame: From the day of CRT and EP procedure until patient discharge, expected stay is an average of 3 days
Measure: Number; unit: ADVERSE EVENTS
Arm/Group | CRT Group | EP Group
Number analyzed (Participants) | 142 | 419
ADVERSE EVENTS | 6 | 12

ADVERSE EVENTS:
Time Frame: The safety surveillance and the safety reporting, both performed by the investigator, started as soon as the subject was enrolled in this study and continued until the last study visit has been completed, i.e. discharge visit, the subject is deceased, or the subject/investigator prematurely withdraws the subject from the study.
Arm/Group | CRT Group | EP Group
All-Cause Mortality (participants affected / at risk) | 0/142 | 0/419
Serious Adverse Events (participants affected / at risk) | 5/142 | 12/419
Other Adverse Events (participants affected / at risk) | 0/142 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRT Group (N=142) | EP Group (N=419)
Arrhyrhmia (Cardiac disorders) | 1 (1) | 2 (2)
Bleeding (non-hematoma) (Vascular disorders) | 1 (1) | 0 (0)
Cardiac Perforation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Tamponade (Cardiac disorders) | 0 (0) | 1 (1)
Coronary Sinus Perforation (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 2 (2)
Phrenic Nerve/Diaphragmatic Stimulation (Nervous system disorders) | 1 (1) | 0 (0)
Pseudoaneurysm (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Stroke (Vascular disorders) | 0 (0) | 2 (2)
Syncope Unknown Etiology (General disorders) | 1 (1) | 0 (0)
OTHER (General disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRT Group (N=142) | EP Group (N=11)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Bleeding(Non-Hematoma) (Vascular disorders) | 0 (0) | 2 (2)
Chest Pain/Discomfort (Cardiac disorders) | 0 (0) | 2 (2)
Hematoma (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
New Or Worsened Angina (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Infections and infestations) | 0 (0) | 1 (1)
Pseudoaneurysm (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thromboembolism (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-04): https://cdn.clinicaltrials.gov/large-docs/12/NCT02470312/Prot_SAP_000.pdf